CLINICAL TRIAL: NCT02824107
Title: INEqualities in Health Psychosocial Determinants of Neuro and Cardio-V@scuLar Disease: Identification of Novel Levers for Secondary Prevention
Brief Title: Psychosocial Risk Factors in Stroke and Myocardial Infarction
Acronym: INEV@L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Béjot PARI 2015
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Myocardial Infarction; Stroke
MeSH Terms: conditions — Myocardial Infarction; Stroke | interventions — Blood Specimen Collection; Surveys and Questionnaires; Psychology

ARMS (2):
- patients with myocardial infarction (Experimental)
  Interventions: Biological: blood sample; Behavioral: questionnaires for psychosocial factors
- patients with stroke (Experimental)
  Interventions: Biological: blood sample; Behavioral: questionnaires for psychosocial factors

INTERVENTIONS:
Biological: blood sample
Behavioral: questionnaires for psychosocial factors

SUMMARY:
The aim of this study is to identify groups of subjects at risk of recurrence in secondary prevention based on Psychosocial Factors.

The aim is also to propose novel levers to reduce health inequalities in this population so as to develop new prevention strategies for neuro- and cardio-vascular health This study is based on data from questionnaires (Quality of life at work, perceived stress, perceived disease severity) and on behavior indicators (factors related to lifestyle: alcohol, smoking, obesity, sedentarity).

Biomarkers of endothelial function (ADMA) will also be assayed. It's an interventional study because of blood sample

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided oral consent to participate
* Patients over 18 years
* Patients hospitalized for type 1 MI or ischemic stroke/TIA < 24H after symptom onset
* Age < 65 years
* With a professional activity (INSEE definition) at the time of the neuro or cardiovascular event
* At least one of the following risk factors: current smoking, obesity (waist circumference > 88 cm (W)/102 cm (M) or a waist/hip ratio 0.85(W)/0.9(M), sedentarity (physical activity < 150 min / week), alcohol consumption (> 3 standard glasses per day for men, > 2 standard glasses/d for women)

Exclusion Criteria:

* Adult under guardianship
* Patients without national health insurance cover
* Pregnant or breast-feeding women
* Clinical state making it impossible to use questionnaires or to measure risk factors
* Stroke or TIA not related to atheroma or cardioembolism (dissection, hemopathy…)
* type > 1 MI

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
number of psychosocial factors (PSF) on the level of risk for neuro-cardiovascular disease. | through the completion study an average of 6 month

SECONDARY OUTCOMES:
study the proportion of diméthyl-arginine asymetrical (ADMA) in patients with PSF | 1st day

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France